CLINICAL TRIAL: NCT03904888
Title: Conventional Versus Robot Assisted Laparoscopic Inguinal Hernia Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, Head of Surgery Department, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Coraline Study
Record Dates: First submitted 2019-03-19; First posted 2019-04-05 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- l-TAPP without local anesthetics (Other): These patients will undergo a laparoscopic surgery without local anaesthetics.
  Interventions: Procedure: l-TAPP
- l-TAPP with local anesthetics (Other): These patients will undergo a laparoscopic surgery with local anaesthetics.
  Interventions: Procedure: l-TAPP; Procedure: local anesthetics
- r-TAPP without local anesthetics (Other): These patients will undergo a robot-assisted surgery without local anaesthetics.
  Interventions: Procedure: r-TAPP
- r-TAPP with local anesthetics (Other): These patients will undergo a robot-assisted surgery with local anaesthetics.
  Interventions: Procedure: r-TAPP; Procedure: local anesthetics

INTERVENTIONS:
Procedure: r-TAPP — Robot-assisted repair
  Arms: r-TAPP with local anesthetics; r-TAPP without local anesthetics
Procedure: l-TAPP — Laporoscopic repair
  Arms: l-TAPP with local anesthetics; l-TAPP without local anesthetics
Procedure: local anesthetics — local anesthetics will be administred
  Arms: l-TAPP with local anesthetics; r-TAPP with local anesthetics

SUMMARY:
Evaluate the early postoperative course of patients undergoing laparoscopic inguinal hernia repair with either a conventional or a robot assisted approach and with or without the injection of the trocar wounds with a local anesthetic.

DETAILED DESCRIPTION:
Introduction Inguinal hernia is a common disease with a high lifetime risk; 27 % for men and 3% for women. These hernias can be categorized as lateral, medial or femoral according to the classification of the European Hernia Society. The manifestations may vary from an asymptomatic swelling till an incarcerated or strangulated hernia requiring an urgent operation.

The introduction of mesh reinforcement for groin hernia repair has resulted in reducing the rate of recurrences and chronic pain. Moreover, laparoscopic repair techniques made it possible to place the mesh in de pre-peritoneal space by a transperitoneal (TAPP) or pre-peritoneal (TEP) approach. These minimally invasive techniques are not only associated with less chronic pain or numbness, but also with an earlier return to normal activities or work. A favor for one of the two techniques has not yet been proven.

At the Hernia Center Maria Middelares a laparoscopic transabdominal pre-peritoneal (l-TAPP) approach is favored in the majority of adult patients presenting with a groin hernia since more than 20 years. The investigators have adopted a technique using one large pre-peritoneal self-fixating mesh that covers both groins in bilateral laparoscopic repairs. In September 2016 the investigators started to use a robot assisted laparoscopic approach (r-TAPP) for groin hernia repair and built proficiency in this technique with 120 cases operated in the first year of adoption. Barriers to adopting robot assisted groin hernia repair are insufficient availability of the robot, perception of longer operative time, perceived lack of clinical benefit for the patient and increased cost for instrumentation.

In a learning curve study using the daVinci Xi robotic system the investigators have shown that after about 25 cases the skin to skin operating time for r-TAPP equals the skin to skin operating time for l-TAPP. Similarly the overall OR time (patient in and out of the OR) is not increased for r-TAPP compared to l-TAPP if the whole team including nurses and anesthetists have become proficient in robotic assisted surgery (Clinical Trials identifier: NCT0975401).

The investigators standard technique for repair of bilateral groin hernias is to use a self-fixating mesh placed in a pre-peritoneal position with a TAPP approach. The investigator prefers to use one large mesh covering the myopectineal orifice of both groins with a width of 28 cm and a length of 13 cm. The mesh used is a Progrip self-fixating mesh (Medtronic, US), which is a monofilament polyester mesh to which resorbable PLA grips have been added to fixate the mesh to the underlying tissue during the period of mesh ingrowth and incorporation. This technique has been studied in our department in a prospective study focusing on early and one year outcome and has shown favorable results (Clinical Trials identifier: NCT02525666 ).

This study aims to differentiate between the early postoperative recovery after laparoscopic repair of bilateral groin hernias treated either with r-TAPP or with l-TAPP.

A total of 200 male and female patients will be entered in the trial in Maria Middelares Ghent, for which an inclusion period of 24 months is anticipated. Patients will be screened and invited to participate at the outpatient clinic.

Study set-up:

* Based on clinical examination and/or ultrasonography 200 patients will be selected.
* Preoperative, during the outpatients' visit, patients will be asked to sign Informed Consent and to fill out the EuraHS-QoL (Quality of Life score) questionnaire.
* Patients will be randomized, to receive either conventional laparoscopic repair (100 patients) or robot assisted laparoscopic repair (100 patients). Patients will be blinded to the surgical method.
* Furthermore patients will be randomized to either receive local anesthetics (50 patients in each group) or none (50 patients in each group)
* Postoperatively, patients will be invited for clinical follow-up with quality of life evaluations with the EuraHS-QoL score at 1 month and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients presenting with a bilateral inguinal hernia planned for a minimal invasive laparoscopic repair

Exclusion Criteria:

* Age below 18 years
* unilateral groin hernia repair
* incarcerated hernias
* open hernia repair
* no informed consent
* pregnant women
* ASA score 4 or more
* patient included in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
change in PADSS score | change of Baseline PADSS score up to 24h after surgery or unitl score is ≥ 9
  Time postoperative for the patient to get fit for discharge as determined by a PADSS score (Post Anesthesia Discharge Scoring System) to reach ≥ 9 (10 is maximum). The score will be taken at 2 hourly intervals after surgery (0 hours,2 hours,4 hours,6 hours,8 hours,10 hours,12 hours,14 hours,16 hours,18 hours,20 hours,22 hours,24 hours) up to 24 hours or unitl score is ≥ 9.

SECONDARY OUTCOMES:
Recurrence rate | at 12 month
  Recurrence rate will be assessed at 12 months post-operatively
Quality of Life assessment: EuraHS Quality of Life questionnaire | 1 month and 12 months post-operatively
  Quality of Life assessment using the EuraHS Quality of Life questionnaire. The questionnaire consists of 9 questions. Each question has a scale from 0-10, wherease 0 is considered the best outcome. Total score (max.90) is assessed by summerizing the scale of each question.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD,PhD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No